CLINICAL TRIAL: NCT05086237
Title: Text Message Follow-up for Patients Who Have Missed Well-Child Visits: Randomized Controlled Trial
Brief Title: Well-Child Visit Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00074978-RCT
Record Dates: First submitted 2021-09-15; First posted 2021-10-20 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-08

CONDITIONS: Child Health; Text Messaging
Keywords: child health; well child visits; text messaging

STUDY DESIGN:
Intervention Model Description: The second phase of the study will be an randomized controlled trial to randomly assign parents/guardians of children who missed a WCV to an intervention condition or no intervention, and assess reasons for missed visits and experiences at last visit. Each reminder message will at minimum direct parents/guardians to reschedule by phone or by the patient portal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reminder (Experimental): Participants will be sent a text message reminder of their missed well-child visit.
  Interventions: Other: Text message reminders
- Treatment as usual (No Intervention): This group will receive treatment as usual, which involves no text messaging follow-up.

INTERVENTIONS:
Other: Text message reminders — Text messages will be sent to parents/guardians of children ages 0 to 17 years who missed their well child visits.
  Arms: Reminder

SUMMARY:
This project will use Twilio as a platform for a text messaging campaign to implement timely follow up with parents/guardians of children ages 0 to 17 years who have missed Well Child Visits (WCVs). The first phase of this project was an open trial. This second phase of the study will be a randomized controlled trial (RCT) to randomly assign parents/guardians of children who missed a WCV to an intervention condition or no intervention, and assess reasons for missed visits and experiences at last visit. Parents/guardians will receive text messages notifying them of missed visits and prompting them to reschedule, as well as inviting them to complete an online survey. Each reminder message will at minimum direct parents/guardians to reschedule by phone or by the patient portal. Outcomes of the follow-up campaign will be evaluated, including rescheduled visits within 6 weeks of missed visit and attendance at rescheduled visit. This aim will incorporate patient Electronic Health Record (EHR) data into mixed effects logistic regressions for the primary study outcomes.

DETAILED DESCRIPTION:
Well-Child visits (WCV) are an opportunity to maximize the health and future well-being and development of children. Missed visits, however, can result in negative outcomes for patients and families and for the healthcare system. For patients, missed primary care visits can result in greater Emergency Department (ED) visits and hospitalizations, and in delays in diagnosing a variety of medical conditions, including identification of child abuse and neglect. For healthcare systems, missed visits result in decreased efficiency, lower quality measures, decreased provider productivity, and loss in revenue. Although smart phones are nearly ubiquitous, even among more economically disadvantaged populations, literature to date has reported only on using text messages for pre-visit reminders. There is a tremendous opportunity to study use of text messaging to engage families in follow-up for missed WCV. Even more so, testing the use of text messages with different content is missing, as well as using text messages to invite patients to share reasons for missing the last WCV.

ELIGIBILITY:
Inclusion Criteria:

Patients included in text messaging campaign (caregivers receive text messages):

* Are 0-17 years
* No-showed for a well-child visit scheduled at one of five locations: Pediatrics-Downtown Health Plaza, Family Medicine-Piedmont Plaza, Pediatrics-Winston East, Family Medicine-Peace Haven, or Pediatrics-Clemmons
* Have a phone number on record for a primary caregiver
* With primary language for contact that is English or Spanish

Caregivers must be 18 years or older

Exclusion Criteria:

Patients who:

* Are 18+ years old
* No-showed for a different type of visit, or no-showed for a WCV at a different practice location
* Already rescheduled their appointment by the time the sample list was generated
* Have primary language specified that is not English or Spanish.

Caregivers who are under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 739 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Number of rescheduled well child visits | 6 weeks after missed well child visit
  If parent/guardian rescheduled well child visit
Number of completed (rescheduled) well child visits | 6 weeks after missed well child visit
  If parent/guardian completed (rescheduled) well child visit

SECONDARY OUTCOMES:
Number of child patient emergency department visits | 6 weeks after missed well child visit
  If child patient had an emergency department visit
Number of child patient hospitalizations | 6 weeks after missed well child visit
  If child patient required hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Poehling, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Debinski B, Daniel SS, Rigdon J, Mayfield A, Tzintzun T, Poehling KA. A Pilot Randomized Controlled Trial of Text Messages to Improve Well-Child Visit Attendance After No-Show. Acad Pediatr. 2024 Nov-Dec;24(8):1210-1219. doi: 10.1016/j.acap.2024.06.003. Epub 2024 Jun 7. PMID 38852906

DOCUMENTS (1):
  • Informed Consent Form (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT05086237/ICF_000.pdf